CLINICAL TRIAL: NCT02413463
Title: Augmented Medial Rectus Muscle Recession Versus Medial Rectus Recession With Posterior Scleral Fixation in Partially Accommodative Esotropia
Brief Title: Augmented Medial Rectus Muscle Recession Versus Posterior Scleral Fixation in Partially Accommodative Esotropia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awadein, Professor of Ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HHH
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Partially Accommodative Esotropia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented recession (Active Comparator): The medial rectus muscle will be exposed and hooked through a limbal approach. The muscle will then be secured with 6-0 polyglactin sutures. The medial rectus muscles will then be recessed using standard tables with the surgical dose targeting the average of the largest and smallest angles
  Interventions: Procedure: augmented recession
- Faden (Active Comparator): Medial rectus muscle recession will be performed as described above with the surgical dose targeting the smallest pre-operative angle. The muscle will then fixated to the sclera using 6/0 polyester sutures placed in a mattress like with the anterior and the posterior sutures passing through both the edge of muscle and the sclera 12 mm and 14 mm from the muscle insertion, respectively.
  Interventions: Procedure: Faden

INTERVENTIONS:
Procedure: augmented recession — medial rectus muscle recession using augmented formula ( average of the distance angle with correction and the near angle without correction)
  Arms: Augmented recession
Procedure: Faden — medial rectus muscle recession (using the distance angle with correction) with posterior scleral fixation( Faden)
  Other Names: Posterior scleral fixation
  Arms: Faden

SUMMARY:
Prospective randomized interventional comparative study

DETAILED DESCRIPTION:
A prospective controlled interventional study will be performed on patients with partially accommodative esotropia. An informed consent for the surgery will be obtained from all patients. All patients' guardians will receive a thorough explanation of the study design and aims, and sign a written informed consent.

An estimation of sample size was performed considering a study power of 0.8 with an alpha error of 0.05 aiming to detect a difference of 5 Δ in the postoperative angle disparity between the 2 groups, assuming a postoperative standard deviation of 6 Δ 9. Based on this estimation, a total of 24 eyes were found to be adequate in each group, and considering a 25% dropout during the follow-up, recruitment of 30 study subjects in each group will be targeted

All patients will receive a full ophthalmological assessment including history taking, measurement of uncorrected and best-corrected visual acuity, cycloplegic refraction, anterior segment examination, as well as a dilated fundus examination.

In addition, all patients will have a detailed motor examination during the initial evaluation and at each follow-up period. The angle of misalignment will be measured by the prism and alternating cover tests for both distance and near with and without glasses. The angle of horizontal misalignment will also be measured in side gazes and in straight up and down gazes. Measurement of the angle of deviation in up and down gazes will be done by tilting the head, approximately 25 degrees down and up respectively, with the patient fixing on a distance target. The difference between the angles of horizontal misalignment in up and down gazes will be used to calculate the amount of pattern strabismus if present.

The ductions and versions in all cardinal directions of gaze will be analyzed before surgery and thereafter during the postoperative follow up visits. Underaction will be measured on a 4-point scale ranging from -1 to -4. Similarly overaction will be measured on a 4-point scale ranging from +1 to +4.

In all patients cycloplegic refraction will be performed using cyclopentolate 1% eye drops instilled 3 times 10 minutes apart with the last time 30 minutes before refraction. Patients with hypermetropia with a spherical equivalent >= +1.5 D will then prescribed the full cycloplegic refraction and then re-evaluated with spectacles one month later. Patients who appear to have a partially accommodative esotropia defined as residual esotropia >8 PD for distance with spectacles will have repeat refraction using atropine 1% drops 3 times a days for 3 days before refraction.

After ensuring that full cycloplegic refraction was prescribed, patients will then evaluated with glasses to identify those with partially accommodative esotropia without convergence excess. Patients will be included in the study if the residual distance angle with cycloplegic prescription was > 15PD. Patients with convergence excess esotropia, defined as the angle of deviation with glasses for near exceeding that for distance by 15 PD or more will be excluded from the study.

Amblyopia, defined as a difference of 0.3 logMAR in verbal children (3 lines on the standard logMAR visual acuity chart) or a strong unilateral fixation preference using an accommodative target in infants and preverbal children will be treated before surgery following the standard clinical practice using part-time occlusion and in concordance with the PEDIG guidelines.

The smallest angle of deviation will be defined as the corrected angle for distance. The largest angle is defined as the angle for near measured without correction. The angle disparity is defined as the difference between the largest and smallest angles.

Patients were randomly allocated using a random table to one of two groups. In one group bilateral augmented MR muscle recession will be performed (augmented group). In the other group bilateral MR muscle recession combined with posterior scleral fixation sutures will be performed (Faden group).

The surgeries were performed using the same surgical technique. In both groups the medial rectus muscle will be exposed and hooked through a limbal approach. The muscle will then secured with 6-0 polyglactin sutures.

In the augmented group, the medial rectus muscles will be recessed using standard tables with the surgical dose targeting the average of the largest and smallest angles.

In the Faden group, medial rectus muscle recession will be performed as described above with the surgical dose targeting the smallest pre-operative angle. The muscle will then be fixated to the sclera using 6/0 polyester sutures placed in a mattress like with the anterior and the posterior sutures passing through both the edge of muscle and the sclera 12 mm and 14 mm from the muscle insertion, respectively.

Patients will be followed up at 1 week, 1 month, 3 months and 6 months after surgery. The distance and near angles of deviation, with and without glasses, and the angle disparity were measured at each follow up visit and the ductions and versions will be assessed in all patients.

Patients will be considered to have successful outcome if both the distance and near angles with spectacles were less than 8 PD esotropia/phoria. Patients who develop any exophoria/tropia, or in whom hyperopic correction needed to be reduced for treatment of a consecutive exotropia will be considered to be unsuccessful. In addition, patients will be further subdivided into 2 groups according to the preoperative angle disparity into those with angle disparity 20 PD or less and those with angle disparity more than 20 PD. The success rate in each subgroup was calculated.

For categorical variables (e.g., gender), percent distribution will be used. For continuous variables (e.g. age, angle of deviation), mean, range and standard deviation will be used. Comparisons between the two groups were done using t-test for independent samples for continuous variables and chi square test for categorical variables. Statistical analysis will be performed with SPSS for Windows (SPSS Inc., Chicago, IL).

.

ELIGIBILITY:
Inclusion Criteria:

* Acquired residual esotropia greater than 14 PD at distance fixation that exists despite full correction of hypermetropic refractive error with the angle of deviation for near not exceeding that of distance by more than 15 PD
* Lack of previous extra ocular muscle surgery

Exclusion Criteria:

* Fully accommodative esotropia, partially accommodative esotropia with convergence excess, non-accommodative esotropia or infantile esotropia
* The presence of neurologic, developmental or ocular structural disorders
* History of previous eye surgery
* Patients requiring simultaneous oblique muscles surgery
* Follow up less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Awadein, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Wright KW, Bruce-Lyle L. Augmented surgery for esotropia associated with high hypermetropia. J Pediatr Ophthalmol Strabismus. 1993 May-Jun;30(3):167-70. doi: 10.3928/0191-3913-19930501-09. PMID 8350226
- [Derived] Al-Hayouti H, Awadein A, Gawdat G, Elhilali H. Augmented medial rectus muscle recession versus medial rectus recession with posterior scleral fixation in partially accommodative esotropia: a randomized clinical trial. J AAPOS. 2020 Oct;24(5):274.e1-274.e7. doi: 10.1016/j.jaapos.2020.05.015. Epub 2020 Oct 7. PMID 33038494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with partially accommodative esotropia were recruited from the strabismus clinic of Pediatric Hospital of Cairo University during the period from January 2015 through December 2016. All patients' guardians received a thorough explanation of the study design and aims, and signed a written informed consent.
Groups:
- Faden: Medial rectus muscle recession will be performed as described as in the augmented recession group with the surgical dose targeting the smallest pre-operative angle. The muscle will then fixated to the sclera using 6/0 polyester sutures placed in a mattress like with the anterior and the posterior sutures passing through both the edge of muscle and the sclera 12 mm and 14 mm from the muscle insertion, respectively.
  Faden: medial rectus muscle recession (using the distance angle with correction) with posterior scleral fixation( Faden)
Period: Overall Study
Arm/Group | Augmented Recession | Faden
Started | 30 | 30
Completed | 25 | 28
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Augmented Recession | Faden | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.6 (2.6) | 5.2 (2.4) | 4.9 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 13 | 14 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Spherical equivalent [Mean (Standard Deviation); unit: Diopters] | 4.91 (1.56) | 4.43 (1.74) | 4.67 (1.71)
Best-corrected visual acuity [Geometric Mean (Standard Deviation); unit: logMAR] | 0.09 (0.06) | 0.11 (0.06) | 0.1 (0.05)
Amblyopia [Count of Participants; unit: Participants] | 10 | 12 | 22
Anisometropia [Count of Participants; unit: Participants] | 11 | 13 | 24
Distance angle of deviation with spectacles [Mean (Standard Deviation); unit: Diopters] | 26 (8) | 21 (6) | 24 (6)
Near angle of deviation with spectacles [Mean (Standard Deviation); unit: Diopters] | 29 (8) | 26 (9) | 28 (8)
Distance angle of deviation without spectacles [Mean (Standard Deviation); unit: Diopters] | 47 (13) | 43 (12) | 45 (12)
Near angle of deviation without spectacles [Mean (Standard Deviation); unit: Diopters] | 50 (12) | 50 (15) | 50 (11)
Angle disparity [Mean (Standard Deviation); unit: Diopters] | 22 (8) | 28 (12) | 25 (9)

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Success rate defined as orthotropia or esotropia ≤ 8 prism diopters with the full hypermetropic correction for near and far without changing the preoperative correction.
Time Frame: six months
Measure: Count of Participants; unit: Participants
Arm/Group | Augmented Recession | Faden
Number analyzed (Participants) | 25 | 28
Participants | 12 | 18
Statistical Analysis 1: Comparison: Augmented Recession vs Faden; An estimation of sample size was performed considering a study power of 0.8 with an alpha error of 0.05 aiming to detect a difference of 5 Δ in the postoperative angle disparity between the 2 groups, assuming a postoperative standard deviation of 6 Δ. Based on this estimation, a total of 24 eyes were found to be adequate in each group, and considering a 25% dropout during the follow-up, recruitment of 30 study subjects in each group was targeted; Test type: Superiority — Chi-square test; p = 0.18, Chi-squared — This is the calculated p-value for the success rate in the Augmented Group Vs. Faden Group

2. Secondary Outcome: Angle of Deviation With Spectacles for Both Distance and Near
Description: The angle of deviation after surgery with full hypermetropic correction
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Augmented Recession | Faden
Number analyzed (Participants) | 25 | 28
Diopters
  Angle of deviation with spectacles for distance | -1 (9) | -3 (7)
  Angle of deviation with spectacles for near | 2 (9) | -1 (7)
Statistical Analysis 1: Comparison: Augmented Recession vs Faden; Test type: Superiority; p = 0.22, t-test, 2 sided — This is the calculated p-value for the postoperative angle of deviation with spectacles for distance in Augmented recession vs. Faden group (First row)

3. Secondary Outcome: Angle of Deviation Without Spectacles for Both Distance and Near
Description: The angle of deviation after surgery without correction for both distance and near
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Augmented Recession | Faden
Number analyzed (Participants) | 25 | 28
Diopters
  Angle of deviation without spectacles for distance | 2 (9) | -1 (7)
  Angle of deviation without spectacles for near | 14 (18) | 6 (9)
Statistical Analysis 1: Comparison: Augmented Recession vs Faden; Test type: Superiority; p = 0.02, t-test, 2 sided — This is the calculated p-value for the postoperative angle of deviation without spectacles for near in Augmented recession vs. Faden group (Second row)

4. Secondary Outcome: Angle Disparity
Description: Difference between largest angle and smallest angle
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Augmented Recession | Faden
Number analyzed (Participants) | 25 | 28
Diopters | 15 (3) | 10 (8)
Statistical Analysis 1: Comparison: Augmented Recession vs Faden; Test type: Superiority; p = 0.03, t-test, 2 sided — This is the calculated p-value for the postoperative angle disparity in the Augmented Group Vs. Faden Group

5. Secondary Outcome: Surgery Time
Description: Time to complete the surgery
Time Frame: Intraoperative time
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Augmented Recession | Faden
Number analyzed (Participants) | 25 | 28
Minutes | 28 (4) | 51 (7)
Statistical Analysis 1: Comparison: Augmented Recession vs Faden; Test type: Superiority; p < 0.01, t-test, 2 sided — This is the calculated p-value for the intraoperative time in the Augmented Group Vs. Faden Group

6. Secondary Outcome: Number of Patients Who Developed Intraoperative and/or Postoperative Complications
Description: Number of patients who developed intraoperative and postoperative complications as scleral perforation, fat prolapse, slipped and lost muscles
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Augmented Recession | Faden
Number analyzed (Participants) | 25 | 28
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Augmented Recession | Faden
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/28
Other Adverse Events (participants affected / at risk) | 0/25 | 0/28

LIMITATIONS AND CAVEATS:
lack of sensory tests and relatively short follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT02413463/Prot_SAP_000.pdf